CLINICAL TRIAL: NCT06845995
Title: The Effects of a Synbiotic Supplement on Metabolic & Cognitive Outcomes and Vitamin D Receptor Variants on Bone Health Among Adults
Brief Title: Effects of a Synbiotic Supplement on Metabolic & Cognitive Outcomes Among Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB2021-1078
Record Dates: First submitted 2024-08-23; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2024-10

CONDITIONS: Older Adults; Bioelectrical Impedance; Appetite Hormones; Metabolic Health; Body Composition Measurement; Cognitive Health
Keywords: Synbiotic supplement; Vitamin D receptor variants; Body composition; Bone health; Metabolic outcomes; Muscle strength; Appetite hormons; Cognitive health

STUDY DESIGN:
Intervention Model Description: Potential subjects will be informed of the study through a study being conducted at Nutrition and Metabolic Health Initiative and at local exercise centers for senior adults and independent living communities by flyers and social media, which will give interested subjects contact information. Once interested subjects communicate with the research team, a research personnel will begin screening process by phone or in-person to see if subject qualifies based on inclusion/exclusion criteria. A research team member will schedule an in-person appointment for subjects that qualify for the study. The research team will ask the subjects to sign a consent form in-person prior to the baseline appointment, Once the consent is signed, random assignment to the study group and data collection will begin.
Who Masked: Participant
Masking Description: Participants will not know if they are taking synbiotic or placebo pill once daily.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Daily placebo: The placebo will be one capsule daily and consists of Microcrystalline Cellulose, Hypromellose, Titanium Dioxide.
- Intervention Group-Receive Synbiotic Supplement (Experimental): Daily synbiotic supplement: The synbiotic supplement (contains both probiotic and prebiotic) that will be used in this study is commercially available; Celebrate Balance. The probiotic will be one capsule daily and consists of lactobacillus acidophilus, Bifidobacterium longum, lactobacillus rhamnosus, and lactobacillus gasser at 28,5 Billion Colony-forming units (CFUs) at manufacture / 15 billion CFUs guaranteed at expiration.
  Interventions: Dietary Supplement: Synbiotic supplement

INTERVENTIONS:
Dietary Supplement: Synbiotic supplement — Daily synbiotic supplement: The synbiotic supplement (contains both probiotic and prebiotic) that will be used in this study is commercially available; Celebrate Balance. The probiotic will be one capsule daily and consists of lactobacillus acidophilus, Bifidobacterium longum, lactobacillus rhamnosus, and lactobacillus gasser at 28,5 Billion CFUs at manufacture / 15 billion CFUs guaranteed at expiration
  Arms: Intervention Group-Receive Synbiotic Supplement

SUMMARY:
The goal of this clinical trial is to investigate the effects of a prebiotic and probiotic supplement on metabolic, cognitive, and muscle health in older adults.

Participants in the study will be older adults who will receive a prebiotic and probiotic supplement containing different strains of Lactobacillus acidophilus, Bifidobacterium longum, Lactobacillus rhamnosus, and Lactobacillus gasseri. The study will collect data at baseline and after 3 months of supplementation to compare the effects on metabolic, cognitive, and muscle health. Additionally, genetic variants associated with vitamin D deficiency and muscle phenotypes will be identified in this population.

DETAILED DESCRIPTION:
Objective one of this research is to determine if there are significant differences in metabolic and muscle health including anthropometrics, biochemical, and muscle quality indices using a prebiotic and probiotic supplement containing different strains of Lactobacillus acidophilus, Bifidobacterium longum, Lactobacillus rhamnosus, and Lactobacillus gasseri in older adults.

There are many physiological changes that occur with aging, which include alterations in the gut microbiota. Gut dysbiosis has also been associated with aging as well as immunity and metabolic alterations such as cardiovascular disease, low-grade inflammation and frailty (Badal et al., 2020). Some studies have shown that probiotics can be a potential therapy to restore the balance of healthy human intestinal function and gut bacterial composition of the gut microbiota because they contain microorganisms naturally found in the human microfiora (Lee et al., 2020). The gut microbiota and its associations with aging are related to clinical and metabolic improvements (Badal et al., 2020). Probiotics and functional foods may have a beneficial effect on the gut by increasing the levels of bifidobacteria or modifying subpopulations of lactobacilli (Ale & Binetti, 2021). The gut microbiota is very important to human metabolism because of its' contribution of enzymes that are not encoded by the human genome, for example, the breakdown of polysaccharides, polyphenols, and synthesis of vitamins (Rowland et al., 2018). It is important to identify the effect that environmental factors, dietary factors (pre and probiotics, etc.), and their combined effect on metabolic and muscle health such as body composition, blood parameters, and muscle quality. Literature shows the benefits of synbiotic (pre and probiotic formula) on several cardiovascular risk factors including lipid and glycemic metabolic parameters in elderly patients (Cicero et al.,2021). However, the optimal timing for supplementation, duration of treatment, as well as the type and dose of the prebiotic and synbiotic to be used needs to be contemplated (Ale & Binetti., 2021).

• Objective two will be to identify variant genes associated with vitamin D deficiency and muscle phenotypes among older adults. Genetic variants for vitamin D deficiency have not been thoroughly studied in older adults. Significant associations have been identified between VDR polymorphism and muscle performance phenotypes although results were conflicting (Pratt et al., 2020). Several allelic variations have been described in the VDR gene, including restriction fragment length polymorphisms, such as Fok1 (C/T) (rs10735810/rs2228570) and Bsm1 (A/G) (rs1544410) (Berry & Hypponen, 2011). This will study the effect of genetic variations on the nutritional requirements of an individual and can provide some prediction to help with prevention as well as contribute to personalized dietary management (Crovesy & Rosado, 2019). It could also lead to improved clarification on the association between vitamin D status and patient outcomes following bariatric surgery (Berry & Hypponen, 2011; Davies et al., 2018).

Objective three will be to identify if there are significant differences in cognitive health including memory, attention, executive functioning, biochemical, and psychomotor skills indices using a prebiotic and probiotic supplement containing different strains of Lactobacillus acidophilus, Bifidobacterium longum, Lactobacillus rhamnosus, and Lactobacillus gasseri in older adults. There are many cognitive changes that occur with aging. Probiotics have been proposed to improve cognitive impairment via the gut-brain axis in patients and experimental animal models (Kim et al, 2021), (Asaoka et al, 2022), (Handajani et al, 2022). However, the beneficial role of synbiotics in brain function of healthy older adults remains unclear (Kim et al, 2021).

Objective one:

Based on 0- to 3-month data collection for baseline and post-intervention physiological outcomes: • What are the differences between basal and 3-month post synbiotic supplementation with regard to the following measurements (biological markers, gut QOL, genetic markers, anthropometric variables).

Based on 3-month supplementation of synbiotics from baseline to 3 months:

Does synbiotic supplementation for 3 months (from baseline to 3rd month) improve gut bacterial functions and gut quality of life in older adults compared to no supplementation?

* If participant report improvement in gut quality of life, are these associated with other physiological indicators of metabolic health (i.e. biological markers, genetic markers, anthropometric variables)?
* Is there an association between improved gut microbiota and gut quality of life and physiological indicators of metabolic health?
* Are any associations observed between improved gut microbiota and biological markers, guts QOL, genetic markers, anthropometric variables?

Objective two:

* What is the prevalence of Vitamin D Receptor (DR) genetic variants in this population?
* Are VDR genetic variants associated with vitamin D deficiency and muscle quality (measured by serum levels, body composition and grip strength)?

Objective three:

Based on 0- to 3-month data collection for baseline and post-intervention physiological outcomes:

What are the differences between basal and 3-month post synbiotic supplementation with regard to the following measurements (biological markers, cognitive function tests, and psychomotor skills)?

Based on 3-month supplementation of synbiotics from baseline to 3 months:

If participant report improvement in gut quality of life, are these associated with other indicators of cognitive health (i.e. biological markers, cognitive function tests, and psychomotor skills)?

Is there an association between improved gut microbiota and gut quality of life and indicators of cognitive health?

Are any associations observed between improved gut microbiota and biological markers, cognitive function tests, and psychomotor skills?

ELIGIBILITY:
Inclusion screening:

* ≥65 years of age
* Male and female
* Physically active as defined by participating in activity beyond baseline activities of daily living (dressing, bathing, toileting, continence, eating, and transferring).

Exclusion screening:

* <65 years of age
* Intake of nicotine, alcohol, and/or drugs such as amphetamines, cocaine, marijuana, and opiates
* Intake of antibiotics or probiotics in the past 3 months
* Intake of medications that might interfere with the study outcomes (e.g. bisphosphonates, steroids, calcitonin, thiazides, glucocorticoids)
* Subjects with hypogonadism, hyperparathyroidism or acute or chronic inflammatory diseases including inflammatory bowel disease, infectious diseases, viral infection, cancer, transplant, renal disorders
* Limited mobility
* Self-reported cognitive dysfunction
* Have heart pacemaker
* People with Type 1 diabetes and Type 2 diabetes taking insulin

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-05-21 (Actual); Primary Completion 2024-07-09 (Actual); Study Completion 2024-07-09 (Actual)

PRIMARY OUTCOMES:
Fecal samples (bacterial diversity) | Baseline and at 3 months
  To assess the differences in gut bacteria diversity after 3 months of supplementation with the synbiotic supplement using the 16S rRNA sequencing analysis method.
Fecal samples (transcriptomics) | Baseline and at 3 months
  To assess the gene expression patterns of microorganisms within the gut, both at baseline and after a three-month supplementation with a synbiotic supplement, the investigators will utilize the NovaSeq 6000 sequencing system method.
Serum Glucagon-like peptide-1 (GLP-1) | Baseline and at 3 months
  To evaluate the levels of appetite hormones, including Glucagon-like peptide-1 (GLP-1) within the serum, both at baseline and after a three-month supplementation with a synbiotic supplement, the investigators will employ the Multiplex 96-well plate assay method.
Serum Interleukin-1beta (IL-1beta) | Baseline and at 3 months
  To evaluate the levels of cytokines, including Interleukin-1beta (IL-1beta) within the serum, both at baseline and after a three-month supplementation with a synbiotic supplement, the investigators will employ the Multiplex 96-well plate assay method.
Serum Noradrenaline/Norepinephrine | Baseline and at 3 months
  To evaluate the serum levels of Noradrenaline/Norepinephrine both at baseline and after a three-month supplementation with a synbiotic supplement. These will be analyzed with ELISA kits.
Serum Vitamin D | Baseline and at 3 months
  To evaluate the levels of vitamin D, within the serum, both at baseline and after a three-month supplementation with a synbiotic supplement. These will be analyzed at a clinical pathology laboratory.
Serum Total Cholesterol | Baseline and at 3 months
  To evaluate the level of total cholesterol within the serum, both at baseline and after a three-month supplementation with a synbiotic supplement. These will be analyzed at a clinical pathology laboratory.
gut quality of life questionnaire | Baseline and at 3 months
  To evaluate the quality of life levels related to gut condition, both at baseline and after three months of supplementation with the synbiotic supplement, the investigators will use the Gut Quality of Life Questionnaire. This is an 11-item questionnaire regarding GI symptoms with a score range of 0 - 44. The lower the score the more negative GI symptoms.
Serum Peptide YY (PYY) | Baseline and at 3 months
  To evaluate the levels of appetite hormones, including Peptide YY (PYY) within the serum, both at baseline and after a three-month supplementation with a synbiotic supplement, the investigators will employ the Multiplex 96-well plate assay method.
Serum Ghrelin | Baseline and at 3 months
  To evaluate the levels of appetite hormones, including ghrelin within the serum, both at baseline and after a three-month supplementation with a synbiotic supplement, the investigators will employ the Multiplex 96-well plate assay method.
Serum Leptin | Baseline and at 3 months
  To evaluate the levels of appetite hormones, including leptin within the serum, both at baseline and after a three-month supplementation with a synbiotic supplement, the investigators will employ the Multiplex 96-well plate assay method.
Serum Insulin | Baseline and at 3 months
  To evaluate the levels of appetite hormones, including insulin within the serum, both at baseline and after a three-month supplementation with a synbiotic supplement, the investigators will employ the Multiplex 96-well plate assay method.
Serum Glucagon | Baseline and at 3 months
  To evaluate the levels of appetite hormones, including glucagon within the serum, both at baseline and after a three-month supplementation with a synbiotic supplement, the investigators will employ the Multiplex 96-well plate assay method.
Serum Tumor Necrosis Factor Alpha (TNF-α) | Baseline and at 3 months
  To evaluate the levels of cytokines, including Tumor Necrosis Factor Alpha (TNF-α) within the serum, both at baseline and after a three-month supplementation with a synbiotic supplement, the investigators will employ the Multiplex 96-well plate assay method.
Serum Interferon gamma (IFNG or IFN-γ) | Baseline and at 3 months
  To evaluate the levels of cytokines, including Interferon gamma (IFNG or IFN-γ) within the serum, both at baseline and after a three-month supplementation with a synbiotic supplement, the investigators will employ the Multiplex 96-well plate assay method.
Serum Interleukin-6 (IL-6) | Baseline and at 3 months
  To evaluate the levels of cytokines, including Interleukin-6 (IL-6) within the serum, both at baseline and after a three-month supplementation with a synbiotic supplement, the investigatorswill employ the Multiplex 96-well plate assay method.
Serum Interleukin-1 receptor (IL-1R) | Baseline and at 3 months
  To evaluate the levels of cytokines, including interleukin-1 receptor (IL-1R) within the serum, both at baseline and after a three-month supplementation with a synbiotic supplement, the investigators will employ the Multiplex 96-well plate assay method.
Serum Interleukin-10 (IL-10) | Baseline and at 3 months
  To evaluate the levels of cytokines, including Interleukin-10 (IL-10) within the serum, both at baseline and after a three-month supplementation with a synbiotic supplement, the investigators will employ the Multiplex 96-well plate assay method.
Serum Dopamine | Baseline and at 3 months
  To evaluate the serum levels of dopamine both at baseline and after a three-month supplementation with a synbiotic supplement. These will be analyzed with ELISA kits.
Serum Serotonin | Baseline and at 3 months
  To evaluate the serum levels of serotonin both at baseline and after a three-month supplementation with a synbiotic supplement. These will be analyzed with ELISA kits.
Serum Brain-derived neurotrophic factor (BDNF) | Baseline and at 3 months
  To evaluate the serum levels of Brain-derived neurotrophic factor (BDNF) both at baseline and after a three-month supplementation with a synbiotic supplement. These will be analyzed with ELISA kits.
Serum Precursor proneurotrophin isoform of BDNF (pro-BDNF) | Baseline and at 3 months
  To evaluate the serum levels of precursor proneurotrophin isoform of BDNF (pro-BDNF) both at baseline and after a three-month supplementation with a synbiotic supplement. These will be analyzed with ELISA kits.
Serum Cortisol | Baseline and at 3 months
  To evaluate the serum levels of Cortisol both at baseline and after a three-month supplementation with a synbiotic supplement. These will be analyzed with ELISA kits.
Serum Insulin-like growth factor-1 (IGF-1) | Baseline and at 3 months
  To evaluate the serum levels of Insulin-like growth factor-1 (IGF-1) both at baseline and after a three-month supplementation with a synbiotic supplement. These will be analyzed with ELISA kits.
Serum LDL cholesterol | Baseline and at 3 months
  To evaluate the levels of LDL cholesterol within the serum, both at baseline and after a three-month supplementation with a synbiotic supplement. These will be analyzed at a clinical pathology laboratory.
Serum Triglycerides | Baseline and at 3 months
  To evaluate the levels of triglycerides within the serum, both at baseline and after a three-month supplementation with a synbiotic supplement. These will be analyzed at a clinical pathology laboratory.
Serum Glucose | Baseline and at 3 months
  To evaluate the levels of glucose within the serum, both at baseline and after a three-month supplementation with a synbiotic supplement. These will be analyzed at a clinical pathology laboratory.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Galyean, Principal Investigator — Texas Tech Nutritional Sciences
Locations (1):
- Shannon Galyean, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available upon request of corresponding author.
Supporting Information: CSR
Time Frame: after publication
Access Criteria: IPD will be available upon request of corresponding author.

REFERENCES:
- [Background] Amit-Romach E, Uni Z, Cheled S, Berkovich Z, Reifen R. Bacterial population and innate immunity-related genes in rat gastrointestinal tract are altered by vitamin A-deficient diet. J Nutr Biochem. 2009 Jan;20(1):70-7. doi: 10.1016/j.jnutbio.2008.01.002. Epub 2008 May 20. PMID 18495461
- [Background] Aron-Wisnewsky J, Prifti E, Belda E, Ichou F, Kayser BD, Dao MC, Verger EO, Hedjazi L, Bouillot JL, Chevallier JM, Pons N, Le Chatelier E, Levenez F, Ehrlich SD, Dore J, Zucker JD, Clement K. Major microbiota dysbiosis in severe obesity: fate after bariatric surgery. Gut. 2019 Jan;68(1):70-82. doi: 10.1136/gutjnl-2018-316103. Epub 2018 Jun 13. PMID 29899081
- [Background] Delzenne NM, Neyrinck AM, Backhed F, Cani PD. Targeting gut microbiota in obesity: effects of prebiotics and probiotics. Nat Rev Endocrinol. 2011 Aug 9;7(11):639-46. doi: 10.1038/nrendo.2011.126. PMID 21826100
- [Background] Delzenne NM, Neyrinck AM, Cani PD. Modulation of the gut microbiota by nutrients with prebiotic properties: consequences for host health in the context of obesity and metabolic syndrome. Microb Cell Fact. 2011 Aug 30;10 Suppl 1(Suppl 1):S10. doi: 10.1186/1475-2859-10-S1-S10. Epub 2011 Aug 30. PMID 21995448
- [Background] Fernandes R, Beserra BT, Mocellin MC, Kuntz MG, da Rosa JS, de Miranda RC, Schreiber CS, Frode TS, Nunes EA, Trindade EB. Effects of Prebiotic and Synbiotic Supplementation on Inflammatory Markers and Anthropometric Indices After Roux-en-Y Gastric Bypass: A Randomized, Triple-blind, Placebo-controlled Pilot Study. J Clin Gastroenterol. 2016 Mar;50(3):208-17. doi: 10.1097/MCG.0000000000000328. PMID 25909598
- [Background] Gill SR, Pop M, Deboy RT, Eckburg PB, Turnbaugh PJ, Samuel BS, Gordon JI, Relman DA, Fraser-Liggett CM, Nelson KE. Metagenomic analysis of the human distal gut microbiome. Science. 2006 Jun 2;312(5778):1355-9. doi: 10.1126/science.1124234. PMID 16741115
- [Background] Graessler J, Qin Y, Zhong H, Zhang J, Licinio J, Wong ML, Xu A, Chavakis T, Bornstein AB, Ehrhart-Bornstein M, Lamounier-Zepter V, Lohmann T, Wolf T, Bornstein SR. Metagenomic sequencing of the human gut microbiome before and after bariatric surgery in obese patients with type 2 diabetes: correlation with inflammatory and metabolic parameters. Pharmacogenomics J. 2013 Dec;13(6):514-22. doi: 10.1038/tpj.2012.43. Epub 2012 Oct 2. PMID 23032991
- [Background] Kong LC, Tap J, Aron-Wisnewsky J, Pelloux V, Basdevant A, Bouillot JL, Zucker JD, Dore J, Clement K. Gut microbiota after gastric bypass in human obesity: increased richness and associations of bacterial genera with adipose tissue genes. Am J Clin Nutr. 2013 Jul;98(1):16-24. doi: 10.3945/ajcn.113.058743. Epub 2013 May 29. PMID 23719559
- [Background] LeBlanc JG, Milani C, de Giori GS, Sesma F, van Sinderen D, Ventura M. Bacteria as vitamin suppliers to their host: a gut microbiota perspective. Curr Opin Biotechnol. 2013 Apr;24(2):160-8. doi: 10.1016/j.copbio.2012.08.005. Epub 2012 Aug 30. PMID 22940212
- [Background] Mondul AM, Weinstein SJ, Albanes D. Vitamins, metabolomics, and prostate cancer. World J Urol. 2017 Jun;35(6):883-893. doi: 10.1007/s00345-016-1878-3. Epub 2016 Jun 23. PMID 27339624
- [Background] Ogden CL, Carroll MD, Kit BK, Flegal KM. Prevalence of childhood and adult obesity in the United States, 2011-2012. JAMA. 2014 Feb 26;311(8):806-14. doi: 10.1001/jama.2014.732. PMID 24570244
- [Background] Peat CM, Kleiman SC, Bulik CM, Carroll IM. The Intestinal Microbiome in Bariatric Surgery Patients. Eur Eat Disord Rev. 2015 Nov;23(6):496-503. doi: 10.1002/erv.2400. Epub 2015 Oct 1. PMID 26426680
- [Background] Rossi M, Amaretti A, Raimondi S. Folate production by probiotic bacteria. Nutrients. 2011 Jan;3(1):118-34. doi: 10.3390/nu3010118. Epub 2011 Jan 18. PMID 22254078
- [Background] Rowland I, Gibson G, Heinken A, Scott K, Swann J, Thiele I, Tuohy K. Gut microbiota functions: metabolism of nutrients and other food components. Eur J Nutr. 2018 Feb;57(1):1-24. doi: 10.1007/s00394-017-1445-8. Epub 2017 Apr 9. PMID 28393285
- [Background] Woodard GA, Encarnacion B, Downey JR, Peraza J, Chong K, Hernandez-Boussard T, Morton JM. Probiotics improve outcomes after Roux-en-Y gastric bypass surgery: a prospective randomized trial. J Gastrointest Surg. 2009 Jul;13(7):1198-204. doi: 10.1007/s11605-009-0891-x. Epub 2009 Apr 18. PMID 19381735
- [Background] Berry D, Hypponen E. Determinants of vitamin D status: focus on genetic variations. Curr Opin Nephrol Hypertens. 2011 Jul;20(4):331-6. doi: 10.1097/MNH.0b013e328346d6ba. PMID 21654390
- [Background] Crovesy L, Rosado EL. Interaction between genes involved in energy intake regulation and diet in obesity. Nutrition. 2019 Nov-Dec;67-68:110547. doi: 10.1016/j.nut.2019.06.027. Epub 2019 Jul 2. PMID 31472367
- [Background] Davies NM, Holmes MV, Davey Smith G. Reading Mendelian randomisation studies: a guide, glossary, and checklist for clinicians. BMJ. 2018 Jul 12;362:k601. doi: 10.1136/bmj.k601. PMID 30002074
- [Background] English WJ, DeMaria EJ, Brethauer SA, Mattar SG, Rosenthal RJ, Morton JM. American Society for Metabolic and Bariatric Surgery estimation of metabolic and bariatric procedures performed in the United States in 2016. Surg Obes Relat Dis. 2018 Mar;14(3):259-263. doi: 10.1016/j.soard.2017.12.013. Epub 2017 Dec 16. PMID 29370995
- [Background] Fallaize R, Macready AL, Butler LT, Ellis JA, Lovegrove JA. An insight into the public acceptance of nutrigenomic-based personalised nutrition. Nutr Res Rev. 2013 Jun;26(1):39-48. doi: 10.1017/S0954422413000024. Epub 2013 Apr 8. PMID 23561449
- [Background] Gemmel K, Santry HP, Prachand VN, Alverdy JC. Vitamin D deficiency in preoperative bariatric surgery patients. Surg Obes Relat Dis. 2009 Jan-Feb;5(1):54-9. doi: 10.1016/j.soard.2008.07.008. Epub 2008 Jul 24. PMID 18848507
- [Background] Moize VL, Pi-Sunyer X, Mochari H, Vidal J. Nutritional pyramid for post-gastric bypass patients. Obes Surg. 2010 Aug;20(8):1133-41. doi: 10.1007/s11695-010-0160-9. PMID 20401543
- [Background] Trovato GM. Behavior, nutrition and lifestyle in a comprehensive health and disease paradigm: skills and knowledge for a predictive, preventive and personalized medicine. EPMA J. 2012 Mar 22;3(1):8. doi: 10.1007/s13167-012-0141-2. PMID 22738244